CLINICAL TRIAL: NCT02472262
Title: Randomized, Single-blinded, Prospective Clinical Trials Comparing the Impact of Legumes vs Corn-soy Flour on Environmental Enteric Dysfunction and Stunting in Rural Malawian Children 6-11 Months
Brief Title: The Impact of Legumes vs Corn-soy Flour on Environmental Enteric Dysfunction in Rural Malawian Children 6-11 Months
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG1
Record Dates: First submitted 2015-06-08; First posted 2015-06-15 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Enteropathy
Keywords: Environmental; Enteric
MeSH Terms: conditions — Intestinal Diseases | interventions — alpha-amylase inhibitor, Phaseolus vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cow pea complementary food (Experimental): A legume-based complementary food made from cowpeas will be given for 6 months,200 kcal/day for children 6-9 months old and 300 kcal/day for children 9-11 months old.
  Interventions: Dietary Supplement: Cow pea complementary food
- Common bean (Experimental): A legume-based complementary food made from common beans will be given for 6 months,200 kcal/day for children 6-9 months old and 300 kcal/day for children 9-11 months old.
  Interventions: Dietary Supplement: Common bean
- Corn Soy Flour (Active Comparator): Corn flour with 10% soy will be given for 6 months, 200 kcal/day for children 6-9 months old and 300 kcal/day for children 9-11 months old.
  Interventions: Dietary Supplement: Corn soy flour

INTERVENTIONS:
Dietary Supplement: Cow pea complementary food — A legume-based complementary food made from cowpeas will be given for 6 months, 200 kcal/day for children 6-9 months old and 300 kcal/day for children 9-11 months old.
  Arms: Cow pea complementary food
Dietary Supplement: Corn soy flour — Corn flour with 10% soy will be given for 6 months, 200 kcal/day for children 6-9 months old and 300 kcal/day for children 9-11 months old.
  Arms: Corn Soy Flour
Dietary Supplement: Common bean — A legume-based complementary food made from common beans will be given for 6 months,200 kcal/day for children 6-9 months old and 300 kcal/day for children 9-11 months old.
  Arms: Common bean

SUMMARY:
To determine if 6 months of legume-based complementary foods is effective in reducing or reversing EED and linear growth faltering in a cohort of Malawian children, aged 6-11 months to see if these improvements are correlated with specific changes in the enteric microbiome.

ELIGIBILITY:
Inclusion Criteria:

children residing in catchment area of Limela, Machinga District and Ntenda (Chikwawa District), Malawi aged 6-11 months youngest eligible child in each household

-

Exclusion Criteria:

Unable to drink 20 mL of sugar water Demonstrating evidence of severe acute malnutrition Apparent need for acute medical treatment for an illness or injury Caregiver refusal to participate and return for 3 and 6 month follow-ups -

-

Ages: 5 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 355 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Manary, MD, Principal Investigator — Washington University School of Medince
Locations (1):
- University of Malawi, Blantyre, Malawi

REFERENCES:
- [Derived] Ordiz MI, Janssen S, Humphrey G, Ackermann G, Stephenson K, Agapova S, Divala O, Kaimila Y, Maleta K, Zhong C, Knight R, Trehan I, Tarr PI, Rusconi B, Manary MJ. The effect of legume supplementation on the gut microbiota in rural Malawian infants aged 6 to 12 months. Am J Clin Nutr. 2020 Apr 1;111(4):884-892. doi: 10.1093/ajcn/nqaa011. PMID 32047925
- [Derived] Ordiz MI, Semba RD, Moaddel R, Rolle-Kampczyk U, von Bergen M, Herberth G, Khadeer M, Roder S, Manary MJ. Serum Amino Acid Concentrations in Infants from Malawi are Associated with Linear Growth. Curr Dev Nutr. 2019 Aug 29;3(10):nzz100. doi: 10.1093/cdn/nzz100. eCollection 2019 Oct. PMID 31620672
- [Derived] Kaimila Y, Pitman RT, Divala O, Hendrixson DT, Stephenson KB, Agapova S, Trehan I, Maleta K, Manary MJ. Development of Acute Malnutrition Despite Nutritional Supplementation in Malawi. J Pediatr Gastroenterol Nutr. 2019 May;68(5):734-737. doi: 10.1097/MPG.0000000000002241. PMID 31022095
- [Derived] Borresen EC, Zhang L, Trehan I, Nealon NJ, Maleta KM, Manary MJ, Ryan EP. The Nutrient and Metabolite Profile of 3 Complementary Legume Foods with Potential to Improve Gut Health in Rural Malawian Children. Curr Dev Nutr. 2017 Sep 21;1(10):e001610. doi: 10.3945/cdn.117.001610. eCollection 2017 Oct. PMID 29955682
- [Derived] Stephenson KB, Agapova SE, Divala O, Kaimila Y, Maleta KM, Thakwalakwa C, Ordiz MI, Trehan I, Manary MJ. Complementary feeding with cowpea reduces growth faltering in rural Malawian infants: a blind, randomized controlled clinical trial. Am J Clin Nutr. 2017 Dec;106(6):1500-1507. doi: 10.3945/ajcn.117.160986. Epub 2017 Nov 1. PMID 29092882
- [Derived] Trehan I, Benzoni NS, Wang AZ, Bollinger LB, Ngoma TN, Chimimba UK, Stephenson KB, Agapova SE, Maleta KM, Manary MJ. Common beans and cowpeas as complementary foods to reduce environmental enteric dysfunction and stunting in Malawian children: study protocol for two randomized controlled trials. Trials. 2015 Nov 14;16:520. doi: 10.1186/s13063-015-1027-0. PMID 26578308

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cow Pea Complementary Food | Common Bean | Corn Soy Flour
Started | 117 | 120 | 118
Completed | 99 | 99 | 93
Not Completed | 18 | 21 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cow Pea Complementary Food | Common Bean | Corn Soy Flour | Total
Number analyzed (Participants) | 117 | 120 | 118 | 355
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 117 | 120 | 118 | 355
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 5.8 (0.3) | 5.8 (0.3) | 5.8 (0.4) | 5.8 (0.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 60 | 53 | 172
  Male | 58 | 60 | 65 | 183
Region of Enrollment [Number; unit: participants]
  Malawi | 117 | 120 | 118 | 355

OUTCOME MEASURES:

1. Primary Outcome: Change in Length-for-age z Score Over 6 Months From Enrollment to End of Study.
Description: Change in length-for-age z score from enrollment to end of study 6 months
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: z-score
Arm/Group | Cow Pea Complementary Food | Common Bean | Corn Soy Flour
Number analyzed (Participants) | 99 | 99 | 93
z-score | -0.14 [-0.24 to -0.04] | -0.27 [-0.38 to -0.16] | -0.27 [-0.35 to -0.19]

2. Primary Outcome: % Lactulose From Dual Sugar Absorption Test at 9 and 12 Months of Age
Description: percent of lactulose found in urine during the dual sugar absorption test
Time Frame: 6 month
Reporting Status: Not Posted, anticipated posting 2020-05

3. Secondary Outcome: 16S Configuration of Fecal Microbiota at 6.5, 7.5, 9, 10.5 and 12 Months of Age Comparing Supplementary Food Groups
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2020-05

4. Secondary Outcome: Mid-upper Arm Circumference at 9 and 12 Months of Age
Description: Mid-upper arm circumference in cm
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2020-05

5. Secondary Outcome: Weight-for-height z Score at 9 and 12 Months of Age
Description: weight for height z-score at 9 and 12 months of age
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2020-05

6. Secondary Outcome: Association of 16S Configuration of Fecal Microbiome With Demographic, Anthropometric, Intestinal Permeability, Sanitation and Antibiotic Exposure Characteristics of the Study Population
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2020-05

ADVERSE EVENTS:
Arm/Group | Cow Pea Complementary Food | Common Bean | Corn Soy Flour
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/120 | 0/118
Other Adverse Events (participants affected / at risk) | 0/117 | 0/120 | 0/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No